CLINICAL TRIAL: NCT05171322
Title: Using Technical Filtering and Clinical Criteria to Reduce Vital Sign Alarms Using Continuous Monitoring in the Ward
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Karoline Kjærgaard, Stud.med, Rigshospitalet, Denmark
Other Study IDs: AWARD (Alert WARD)
Record Dates: First submitted 2021-12-10; First posted 2021-12-28 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Vital Signs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- All patients: All patients included were set up with the WARD monitoring devices.
  Interventions: Device: WARD

INTERVENTIONS:
Device: WARD — The following monitoring devices are included in the WARD monitoring system (as intervention):
  Isansys Life Touch patch: Measures heart rate (HR), respiratory rate (RR) and electrocardiogram (ECG)
  Wearable, wireless Pulse Oximeter (Model 3150 WristOx from Nonin): Measures peripheral oxygen saturation of arterial hemoglobin (SpO2) and pulse rate (PR)
  Blood pressure monitor (Meditech BlueBP-05): Measures BP every 30 minutes during daytime and every 60 minutes during the night
  All included patients are set up with the monitoring devices after surgery when they are back at their ward (with a maximum of 24 hours postoperative). Afterwards they wear the devices for up to 5 days. All measurements are sent through bluetooth to a tablet serving as a gateway which in turn sends data to a central server where the algorithmic processing ensures.

SUMMARY:
The purpose of this study is to describe the extent of vital sign threshold alarm reduction in relation to several simple multilevel minimum duration criteria and artefact removal. We hypothesize that the amount off false alarms will be decreased using different filters.

DETAILED DESCRIPTION:
Introduction: Early identification of patients who are at risk of severe vital sign deterioration is essential in reducing mortality in critically ill patients. Abnormal physiology often precedes adverse outcomes like unexpected cardiac arrest, unexpected admission to intensive care units (ICU) and unexpected death among hospitalized patients.

The system, which is currently being used at Danish hospitals for monitoring patient's vital signs, is the EWS system (Early Warning Score) carried out primarily by nurses. The EWS monitors 7 parameters: Blood pressure (BP), heart rate (HR), blood saturation (SpO2), respiratory rate (RR), temperature, level of alertness and oxygen supplementation. Depending on the measured values, the EWS system determines the intervals with which nurses must measure vital signs. In case of aberrant signs medical staff is informed.

While simple continuous monitoring is rarely used outside the PACU or ICU, it presents the possibility of detecting early signs of deteriorations (ESODs), but has shown to induce alarm fatigue among hospital staff, thus increasing the risk of mortality. In addition the system is based on a "better-safe-than-sorry-logic", where a large amount of false alarms are accepted, rather than risking missing one correct alarm.

Aim: The aim of this study is to describe the extent of vital sign threshold alarm reduction in relation to several simple multilevel minimum duration criteria and artefact removal. We hypothesize that the amount off false alarms will be decreased using different filters.

Methods: The study is a prospective, descriptive cohort study, where patients were included from prospective WARD studies. Data will be analysed using different filters and a duration criteria. First data is analysed without artefact removal, where alarms are collected as in the ward, where alarms are activated if any vitals sign is below or above the threshold for a minimum of 15 seconds. Next data is filtered and analysed with artefact removal and finally data is filtered and analysed with a duration criteria. Furthermore, the available data are without staff interventions and may thus represent cases where the first alert would result in effective treatment and that subsequent alerts were averted. To assess this the data will be analysed for number of alerts if the first alert removed 100%, 75%, 50%, 25% and 0% of the following same alerts within the first hour, the following 3, 6, 12 and 24 hours.

Results: The primary analysis will be number of vital sign threshold alarms/patients/day for the alarms with artefact removal but without a duration criteria compared to the alarms with artefact removal and a duration criteria. The two filters will be compared using either a paired Student's t-test or a paired Mann-Whitney U test. The secondary and tertiary analysis of the secondary and tertiary outcomes will be performed using either a paired Student's t-test or a paired Mann-Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

WARD COPD project (NCT03660501):

* ≥18 years
* Patients admitted to emergency departments or pulmonary wards with AECOPD as admission diagnosis with suspected acute exacerbation of COPD
* The diagnosis had to be sustained in the patient record at the time of inclusion
* Expected admittance longer than 24 hours
* Possibility of an investigator to include the patient within 24 hours from admission

The WARD surgery project (NCT03491137):

* ≥ 60 years
* Elective major abdominal cancer surgery
* Estimated surgical duration ≥ 2 hours.

WARD VASC project (NCT04628858):

* ≥ 18 years
* Patients with PAD which must undergo an open intraligamentary revascularization incl. a. femoralis TEA and intraligamentary bypass
* Patients admitted at the department of vascular surgery 3111 at Rigshospitalet regarding elective surgery
* Patients admitted the day before surgery and have an expected admitting time lasting more than 2 days (postoperatively)

WARD CGM (NCT04473001):

* Adult patients ≥ 18 years
* Patients admitted at Rigshospitalet or Bispebjerg hospital for major abdominal surgery or major orthopedic surgery or major arterial vascular surgery
* Estimated duration of surgery ≥ 1 hour and at least one expected overnight stay at the hospital postoperatively
* Type 1 diabetes or type 2 diabetes treated with insulin or type 2 diabetes treated with oral antihyperglycemic drugs/GLP-1 analogs or patients with no diabetes

Exclusion Criteria:

WARD COPD project (NCT03660501):

* Patients who were not expected to cooperate to wear the monitoring equipment
* Unable to give informed consent
* Patients who were withheld active treatment
* Implanted cardioverter defibrillator or pacemaker
* Severe allergy for plaster/silicone

WARD CODP pilot project (NCT03467815):

* ≥ 18 years
* Patients admitted with AECOPD as admission diagnosis (this diagnosis had to be maintained in the patient record at time of inclusion)

The WARD surgery project (NCT03491137):

* Implanted cardioverter defibrillator or pacemaker
* Allergy to study devices
* Severe cognitive impairment assessed by MMSE
* Inability to cooperate wearing the wireless monitoring equipment

WARD CODP pilot project (NCT03467815):

* Unable to give informed consent
* Inability to cooperate to wear the monitoring equipment
* Active therapy withdrawn
* Expected duration of admission less than 24 hours after possible enrolment
* Allergies to plaster, plastic or silicone

WARD VASC project (NCT04628858):

* Inability to cooperate wearing the wireless monitoring equipment
* Unable to give informed consent due to dementia or other reason.
* Severe allergy for plaster/silicone
* Implanted cardioverter defibrillator or pacemaker
* Patients not expected to be admitted for over 24 hours from possible inclusion time
* Isolated patients/patients with possible MRSA
* Patients who where withheld active treatment
* Patients formerly included in WARD surgery or WARD COPD studies
* Patients with a difference in systolic BP > 20 mmHg between their two arms

WARD CGM (NCT04473001):

* Patients expected not to corporate with study procedures
* Patients allergic to plaster or silicone
* Patients with impaired cognitive function
* Patients with any treatment limitation
* Previous or currently scheduled for pancreatectomy
* Patients with pacemaker or ICD device

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients are included from prospective WARD studies. The WARD surgery project (NCT03491137), the WARD COPD project (NCT03660501), the WARD CGM (NCT04473001), the WARD CODP pilot project (NCT03467815) and the WARD VASC project (NCT04628858).
Sampling Method: Non-Probability Sample
Enrollment: 850 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Calculated number of any vital sign threshold alarms/patient/24 hours (bradypnea, tachypnea, desaturation, sinus tachycardia, bradycardia, hypotension and hypertension). | 24 hours

SECONDARY OUTCOMES:
Number of bradypnea threshold alarms/patient/24 hours. | 24 hours
Number of tachypnea threshold alarms/patient/24 hours. | 24 hours
Number of desaturation threshold alarms/patient/24 hours. | 24 hours
Number of sinus tachycardia threshold alarms/patient/24 hours. | 24 hours
Number of bradycardia threshold alarms/patient/24 hours. | 24 hours
Number of hypotension threshold alarms/patient/24 hours. | 24 hours
Number of hypertension threshold alarms/patient/24 hours. | 24 hours

OTHER OUTCOMES:
Number of vital sign threshold alarms/patient for efficiency levels at 0%, 25%, 50%, 75% and 100%, firstly within the first hour, afterwards following the first 3 hours, 6 hours, 12 hours and 24 hours. | 1 hour, 3 hours, 6 hours, 12 hours and 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Department of Anesthesiology, Centre for Cancer and Organ Diseases, Copenhagen, Copenhagen Ø, Denmark